CLINICAL TRIAL: NCT00447733
Title: Effects of Integrated Treatment to Persons With Mental Disorders and Co-occurring Substance Use Disorders
Brief Title: Integrated Treatment to Persons With Mental Disorders and Co-occurring Substance Use Disorders
Acronym: ROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: SINTEF Health Research (Other)
Responsible Party: Principal Investigator, Rolf W. Grawe, Ph.d.; Assistent Professor; University of Oslo, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 78i068; NFR175394/V50 (Other Grant/Funding Number: The Norwegian Research Council/NFR175394/V50)
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Anxiety Disorders; Mood Disorders; Substance Use Disorders
Keywords: mental health; substance use; treatment
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Substance-Related Disorders; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated treatment (Experimental): Evidence-based psychosocial and pharmacological treatment of both the substance use disorder and the mental health disorder is provided at the same time and by the same therapists in a comprehensive way.
  Interventions: Behavioral: Integrated mental health and substance use treatment
- Treatment as usual (Active Comparator): Non-manualized clinic-based treatment provided by therapists without formal training in integrated treatment of co-occurring disorders.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Integrated mental health and substance use treatment — Psychosocial and drug treatment targeting both the substance use disorder and the psychiatric disorder in an integrated and comprehensive way.
  Other Names: dual disorder treatment; co-occurring disorders
  Arms: Integrated treatment
Behavioral: Treatment as usual — Non-standardized psychiatric outpatient treatment
  Other Names: TAU; non-manualized
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to determine whether Integrated Treatment is effective in the treatment of anxiety and/or depression with co-occurring substance use disorders.

DETAILED DESCRIPTION:
Patients with mental disorders and co-occuring substance use disorders are characterized by high suicide rates, high treatment drop-out rates and long-lasting interpersonal, work, school, health and legal problems. Because mental disorders and substance use disorders co-exist and interact, it may be important to provide a treatment that addresses the substance misuse and mental health problems in an integrated and comprehensive way. Additionally, the health services for patients with mental health and substance use disorders are usually provided by different services and health professionals that rarely cooperate or have qualifications on both kinds of disorders. This also calls for an integration of the services on an organizational level. This approach of integrating services and treatment approaches for both diseases in a comprehensive way is called Integrated Treatment. Several studies have shown that Integrated Treatment is effective in treating the comorbidity of severe mental illness and substance use disorders. The over-all aim of this study is to evaluate the effects of evidence-based Integrated Treatment in anxiety and/or depression with co-occurring substance use disorders. The effects of the treatment will be assesses on changes in substance use and psychopathology.

Comparison: patients receiving treatment-as-usual or non-manualized treatment at general mental health outpatients clinics.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of substance use disorder
* clinical diagnosis of anxiety disorders
* clinical diagnosis of nonpsychotic mood disorders
* written consent
* planning to live in the catchment area during the treatment

Exclusion Criteria:

* schizophrenia spectrum disorders
* other psychotic disorders
* mental retardation
* nicotine abuse/dependency only
* prescription drug abuse/dependency only
* planning to move out of the catchment area during the study
* not able to read or write Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The Symptom Check List 90 (SCL90-r), The Alcohol Use Disorder Identification Test (AUDIT), The Drug Use Disorder Identification Test (DUDIT). | Change during 6 and 12 months follow-up
  We use the SCL-90r to measure symptoms in regard to anxiety, depression and the General Severity Index.
  We use the AUDIT and the DUDIT to measure changes in the use of alcohol and illegal drugs respectively.

SECONDARY OUTCOMES:
The Addiction Severity Index (Europ ASI) | Change during 6 and 12 months follow up
  The Addiction Severity Index (Europ ASI) is used to assess changes in the use of alcohol and illegal substances during the course of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf W. Gråwe, Ph.D, Principal Investigator — Alcohol and Drug Treatment Health Trust in Central Norway; Norwegian Centre of Addiction Research, University of Oslo

REFERENCES:
- [Derived] Wusthoff LE, Waal H, Grawe RW. The effectiveness of integrated treatment in patients with substance use disorders co-occurring with anxiety and/or depression--a group randomized trial. BMC Psychiatry. 2014 Mar 5;14:67. doi: 10.1186/1471-244X-14-67. PMID 24597469
- [Derived] Wusthoff LE, Waal H, Grawe RW. When research meets reality-lessons learned from a pragmatic multisite group-randomized clinical trial on psychosocial interventions in the psychiatric and addiction field. Subst Abuse. 2012;6:95-106. doi: 10.4137/SART.S9245. Epub 2012 Aug 16. PMID 22933843